CLINICAL TRIAL: NCT03708458
Title: Comparative Evaluation of Standard Prophylaxis Versus Divided-dose NSAIDs or Hybrid NSAID and N-acetylcysteine Therapy for the Prevention of Post-ERCP Pancreatitis
Brief Title: Pharmacological Prophylaxis of Post- Endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, PAVEL LAURA, Principal Investigator, PhD Student, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEP_2017
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Post-ERCP Pancreatitis
Keywords: endoscopic retrograde cholangiopancreatography (ERCP); post-ERCP pancreatitis (PEP); Nonsteroidal anti-inflammatory drugs (NSAID's); acetylcysteine (ACC)
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Control group - patients receiving 100 mg indomethacin suppository immediately post ERCP
  Interventions: Drug: indomethacin suppository
- Group A (Active Comparator): Group A - patients receiving N-acetylcysteine (NAC) 600 mg before performing ERCP and indomethacin suppository 50 mg before and after performing ERCP
  Interventions: Drug: indomethacin suppository; Drug: N-acetylcysteine (NAC)
- Group B (Active Comparator): Group B - patients receiving indomethacin suppository 50 mg before and 50 mg after ERCP
  Interventions: Drug: indomethacin suppository

INTERVENTIONS:
Drug: indomethacin suppository — the investigators aimed to perform a comparative study, evaluating the efficacy of three prophylactic approaches aiming to reduce the risk of PEP, using indomethacin and/or N-acetylcysteine -NAC, in different regimens
Drug: N-acetylcysteine (NAC) — the investigators aimed to perform a comparative study, evaluating the efficacy of three prophylactic approaches aiming to reduce the risk of PEP, using indomethacin and/or N-acetylcysteine -NAC, in different regimens
  Arms: Group A

SUMMARY:
The investigators aimed to perform a comparative study, evaluating the efficacy of three prophylactic approaches aiming to reduce the risk of post-ERCP pancreatitis, using pharmacologic agents with different mechanisms of action (NSAIDs and/or acetylcysteine) in three different regimens.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older
* diagnosis of choledocholithiasis
* indication for ERCP procedures
* willingness to participate in the study
* the ability to sign the informed consent

Exclusion Criteria:

* presence of acute pancreatitis or other inflammatory diseases at admission
* pregnancy
* contraindication for NSAID administration
* recent episode of upper digestive bleeding (less than one month)
* hypersensibility to antioxidants hypersensibility to antioxidants
* the necessity of a prophylactic pancreatic stent insertion
* patients' disapproval to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients who develop post ERCP pancreatitis | 24 hours post ERCP
  Comparing and evaluating the efficacy of three pharmacological combination therapies (Indomethacin +/- N-acetylcysteine), aiming to prevent acute post ERCP pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: GHEORGHE BALAN, PhD, Professor, Study Director — "GRIGORE T. POPA" UNIVERSITY OF MEDICINE AND PHARMACY IAŞI
Locations (1):
- Institute of Gastroenterology and Hepatology - St. Spiridon County Clinical Emergency Hospital of Iași, Iași, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dumonceau JM, Andriulli A, Elmunzer BJ, Mariani A, Meister T, Deviere J, Marek T, Baron TH, Hassan C, Testoni PA, Kapral C; European Society of Gastrointestinal Endoscopy. Prophylaxis of post-ERCP pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - updated June 2014. Endoscopy. 2014 Sep;46(9):799-815. doi: 10.1055/s-0034-1377875. Epub 2014 Aug 22. PMID 25148137
- [Background] Yaghoobi M, Rolland S, Waschke KA, McNabb-Baltar J, Martel M, Bijarchi R, Szego P, Barkun AN. Meta-analysis: rectal indomethacin for the prevention of post-ERCP pancreatitis. Aliment Pharmacol Ther. 2013 Nov;38(9):995-1001. doi: 10.1111/apt.12488. Epub 2013 Sep 16. PMID 24099466
- [Background] Levenick JM, Gordon SR, Fadden LL, Levy LC, Rockacy MJ, Hyder SM, Lacy BE, Bensen SP, Parr DD, Gardner TB. Rectal Indomethacin Does Not Prevent Post-ERCP Pancreatitis in Consecutive Patients. Gastroenterology. 2016 Apr;150(4):911-7; quiz e19. doi: 10.1053/j.gastro.2015.12.040. Epub 2016 Jan 9. PMID 26775631
- [Background] Gooshe M, Abdolghaffari AH, Nikfar S, Mahdaviani P, Abdollahi M. Antioxidant therapy in acute, chronic and post-endoscopic retrograde cholangiopancreatography pancreatitis: An updated systematic review and meta-analysis. World J Gastroenterol. 2015 Aug 14;21(30):9189-208. doi: 10.3748/wjg.v21.i30.9189. PMID 26290647
- [Background] Fuentes-Orozco C, Davalos-Cobian C, Garcia-Correa J, Ambriz-Gonzalez G, Macias-Amezcua MD, Garcia-Renteria J, Rendon-Felix J, Chavez-Tostado M, Cuesta-Marquez LA, Alvarez-Villasenor AS, Cortes-Flores AO, Gonzalez-Ojeda A. Antioxidant drugs to prevent post-endoscopic retrograde cholangiopancreatography pancreatitis: What does evidence suggest? World J Gastroenterol. 2015 Jun 7;21(21):6745-53. doi: 10.3748/wjg.v21.i21.6745. PMID 26074713
- [Background] Katsinelos P, Kountouras J, Paroutoglou G, Beltsis A, Mimidis K, Zavos C. Intravenous N-acetylcysteine does not prevent post-ERCP pancreatitis. Gastrointest Endosc. 2005 Jul;62(1):105-11. doi: 10.1016/s0016-5107(05)01574-9. PMID 15990827
- [Background] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Background] Luo H, Zhao L, Leung J, Zhang R, Liu Z, Wang X, Wang B, Nie Z, Lei T, Li X, Zhou W, Zhang L, Wang Q, Li M, Zhou Y, Liu Q, Sun H, Wang Z, Liang S, Guo X, Tao Q, Wu K, Pan Y, Guo X, Fan D. Routine pre-procedural rectal indometacin versus selective post-procedural rectal indometacin to prevent pancreatitis in patients undergoing endoscopic retrograde cholangiopancreatography: a multicentre, single-blinded, randomised controlled trial. Lancet. 2016 Jun 4;387(10035):2293-2301. doi: 10.1016/S0140-6736(16)30310-5. Epub 2016 Apr 28. PMID 27133971